CLINICAL TRIAL: NCT03544840
Title: An Investigation of Trunk Control in Young Children With Down Syndrome
Brief Title: Investigating Trunk Control in Young Children With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Collaborators: American Physical Therapy Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20067
Record Dates: First submitted 2018-05-11; First posted 2018-06-04 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Down Syndrome; Gross Motor Development Delay
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dynamic Standing Device (Experimental): Home program using the Upsee
  Interventions: Other: Physical Therapy Home Program

INTERVENTIONS:
Other: Physical Therapy Home Program — On the first day of the intervention phase (B), the PI will deliver the dynamic standing home program device (Upsee) to the parent and child. The PI will provide training and education to the parent on the device and home program. At the weekly visit to score outcome measures, the PI will check the fit of the devices, ensure compliance, and answer any questions about the home program. Parents will be encouraged to use the device with their child 5 days per week, 30 minutes per day. Parents will keep a daily log sheet to record duration of device use, activities performed, and subjective observations of the child during the intervention (Appendix K). The PI will collect these log sheets each week. The baseline phases (A1 and A2) will last 4 weeks and the intervention phase (B) will last 6 weeks. Part 2 of the study is expected to last 14 weeks.

SUMMARY:
Overall, the purpose of this dissertation research is to investigate trunk control in young children with DS. This will be done in three studies:

1. The purpose of the first study is to determine the reliability of the SATCo in young children with DS. The hypothesis is that the SATCo will demonstrate good (κ > 0.8) interrater and intrarater reliability.
2. The purpose of the second study is to examine the validity of the SATCo with the GMFM-66 and determine whether age and SATCo score predict GMFM-66 score in young children with DS. The hypotheses are that 1) the SATCo will show concurrent validity with the GMFM-66, and 2) both age and SATCo scores will be significant predictors of GMFM-66 scores.
3. The purpose of the third study is to explore the impact of a dynamic standing device (Upsee) on trunk control and motor skills in young children with DS. The hypothesis is that participants will demonstrate a greater change in scores on the SATCo and the GMFM during the dynamic standing home program phase than during the baseline phases.

DETAILED DESCRIPTION:
Literature suggests there is a need to identify effective home programs to supplement physical therapy and improve gross motor function in children with Down syndrome (DS). To study the impact of home programs, effective tools must be employed to measure the incremental changes that occur in young children with DS, both at the body structure and function level and the activity level of the World Health Organization's International Classification of Functioning, Disability and Health (ICF). The Gross Motor Function Measure (GMFM-66) is an effective measure of motor skills at the activity level of the ICF for children with DS; however, there is a lack of sound outcome measures of trunk control for young children with DS. The Segmental Assessment of Trunk Control (SATCo) may be an effective tool for this purpose but has not been studied in this population.

In addition to assessing trunk control in children with DS, intervention strategies for improving trunk control in this population must be investigated. A home program using upright mobility through treadmill training has proven to be effective in accelerating the acquisition of motor skills in infants with DS; however, alternative forms of upright mobility that are more affordable and less cumbersome are needed. The Upsee (Firefly by Leckey, Lisburn, Northern Ireland) shows promise as a dynamic standing device that can be used at home by the parent and child to promote upright mobility. This device has not been studied in young children with DS.

Overall, the purpose of this dissertation research is to investigate trunk control in young children with DS. This will be done in three studies:

1. The purpose of the first study is to determine the reliability of the SATCo in young children with DS. The hypothesis is that the SATCo will demonstrate good (κ > 0.8) interrater and intrarater reliability.
2. The purpose of the second study is to examine the validity of the SATCo with the GMFM-66 and determine whether age and SATCo score predict GMFM-66 score in young children with DS. The hypotheses are that 1) the SATCo will show concurrent validity with the GMFM-66, and 2) both age and SATCo scores will be significant predictors of GMFM-66 scores.
3. The purpose of the third study is to explore the impact of a dynamic standing device (Upsee) on trunk control and motor skills in young children with DS. The hypothesis is that participants will demonstrate a greater change in scores on the SATCo and the GMFM during the dynamic standing home program phase than during the baseline phases.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of DS. This is the diagnosis that is being investigated
2. Speak English. This is the language spoken by the PI.
3. Medically stable, without physician- ordered restrictions. Some children with DS have cardiac surgery or other complications that would contraindicate handling or movement. These children would not be considered medically stable.
4. Between the age of 6 to 24 months. This captures the full range of the outcome measure being investigated.

Exclusion Criteria:

1. Meet inclusion and exclusion criteria for part 1 of the study. Children for part 2 of the study will be a sub-sample of those in part 1 of the study.
2. Between the age of 9 to 18 months. This captures the age when most children with DS are able to bear weight through their lower extremities, but before they can walk independently. This is necessary to be able to use the home programs and demonstrate gross motor changes.
3. Unable to ambulate independently. Children who can walk independently cannot use the home program devices.

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Segmental Assessment of Trunk Control | 20 minutes
  Assesses seated trunk control in children with neuromotor disorders.
Gross Motor Function Measure | 40 minutes
  Assesses gross motor skills in children with Down syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Megan Flores, MPT, Principal Investigator — Student
Locations (1):
- University of St. Augustine for Health Sciences, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ulrich DA, Ulrich BD, Angulo-Kinzler RM, Yun J. Treadmill training of infants with Down syndrome: evidence-based developmental outcomes. Pediatrics. 2001 Nov;108(5):E84. doi: 10.1542/peds.108.5.e84. PMID 11694668
- [Background] Russell D, Palisano R, Walter S, Rosenbaum P, Gemus M, Gowland C, Galuppi B, Lane M. Evaluating motor function in children with Down syndrome: validity of the GMFM. Dev Med Child Neurol. 1998 Oct;40(10):693-701. doi: 10.1111/j.1469-8749.1998.tb12330.x. PMID 9851239
- [Background] Butler PB, Saavedra S, Sofranac M, Jarvis SE, Woollacott MH. Refinement, reliability, and validity of the segmental assessment of trunk control. Pediatr Phys Ther. 2010 Fall;22(3):246-57. doi: 10.1097/PEP.0b013e3181e69490. PMID 20699770
- [Background] Ulrich BD. Opportunities for early intervention based on theory, basic neuroscience, and clinical science. Phys Ther. 2010 Dec;90(12):1868-80. doi: 10.2522/ptj.20100040. Epub 2010 Oct 21. PMID 20966210